CLINICAL TRIAL: NCT03767426
Title: The Effect of Sleep Deprivation and Recovery Sleep on Emotional Memory and Affective Reactivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston College (Other)
Responsible Party: Principal Investigator, Robert Stickgold, Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TC-1
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sleep Deprivation; Sleep
Keywords: Emotion; Memory; Sleep; Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Independent group comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Overnight sleep (No Intervention): Subjects are permitted a night of polysomnograph-recorded sleep before participating in training and testing sessions the next day
- Sleep deprivation (Active Comparator): Subjects sleep deprived before participating in training and testing sessions the next day
  Interventions: Behavioral: Sleep Deprivation
- Daytime Nap (Experimental): Subjects are trained and then retested after a daytime nap
  Interventions: Behavioral: Sleep Deprivation; Behavioral: Daytime nap

INTERVENTIONS:
Behavioral: Sleep Deprivation — Subjects are sleep deprived for an entire night
  Arms: Daytime Nap; Sleep deprivation
Behavioral: Daytime nap — After a night of sleep deprivation, participants will be given a 2 hour nap opportunity
  Arms: Daytime Nap

SUMMARY:
To further understand the impact of acute sleep deprivation and recovery sleep on the processing of emotional information the investigators will address and attempt to answer three questions, (i) how both undisturbed sleep and sleep deprivation affect the processing and retrieval of emotional information, (ii) what neural and psychophysiological mechanisms are associated with these behavioral effects, and (iii) to explore the ability of recovery sleep to reverse the effects of sleep deprivation. Together, these studies will provide a greater breadth and depth of knowledge concerning sleep's role in emotion processing and regulation. Given the growing societal tendency to view sleep as unproductive-foregoing it to lengthen work days and increase social opportunities- such knowledge would be of practical importance for understanding the role of sleep in healthy emotional functioning, particular for individuals experiencing periods of increased stress and emotional distress (e.g., new parents, hospital staff, or combat troops).

DETAILED DESCRIPTION:
Goal 1: How does sleep deprivation impact emotion perception and memory processing? The investigators are interested in how an acute loss of sleep impairs our ability to properly perceive, consolidate, and retrieve emotional information. There has been research on the effect of sleep deprivation on broad areas of cognition, such as attention, working memory, and reasoning ability, but the impact of sleep loss on emotional processing and regulation remains largely unexplored. The investigators aim to characterize how sleep deprivation compared to undisturbed sleep affects the ability to accurately perceive emotion, how it alters the intensity with which emotions are perceived, and the effect that these changes have on the subsequent consolidation and memory retrieval for emotional compared to neutral information.

Goal 2: How are these changes reflected in the neural signal and with psychophysiological measures? The investigators will utilize functional magnetic resonance imaging (fMRI) and measures of autonomic reactivity (heart rate and skin conductance) to characterize the neural and psychophysiological mechanisms underlying these behavioral changes following sleep deprivation compared to a normal night of sleep. This will allow us to pinpoint the brain regions involved in changes following sleep deprivation, and associate these changes with effects on downstream physiological responses.

Goal 3: Can a nap after sleep deprivation restore normal processing of emotional memory and rescue the neural and autonomic markers of sleep deprivation? The investigators are interested in determining if a brief period of recovery sleep is enough to combat the behavioral, neural, and autonomic effects of acute sleep loss, thus a portion of the sleep-deprived participants will be given a 2-hour nap opportunity to quantify its restorative effects. Such information would form the foundation for future research extending and translating these findings into effective sleep-based interventions for healthy and clinical populations alike.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to follow the protocol
* willing and able to meet inclusion criteria for fMRI scanning
* willing to refrain from alcohol and recreational drugs for the duration of the protocol
* normal or corrected to normal vision is required

Exclusion Criteria:

* self-reported sleep disturbances
* left-handedness or ambidexterity
* a history of mental illness or neurological disorder
* the use of any drugs that could affect either sleep or cognitive functioning (e.g., sleeping pills or antidepressants)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphed Face Accuracy and Intensity | 1-24 hours
  Participants are asked to identify and rate emotional intensity of ambiguous emotional faces (happy, sad, angry) that have been morphed with neutral faces. Scores for each emotional domain will be calculated as (i) accuracy score (number of faces correctly identified over total faces seen), and (ii) average emotional intensity rating. Task will be completed at baseline, post-sleep/sleep deprivation, and post-nap/no nap, and within-subject comparisons will determine how interventions impact emotional perception.
Emotional Memory Tradeoff Memory Score | 12-24 hours
  Following sleep or sleep deprivation, participants will complete emotional memory tradeoff recognition task at two time points, separated by a nap or wakefulness. Corrected hit rate will be calculated for negative and neutral scene components as the percentage of correctly identified "old" objects/backgrounds minus percentage of false alarms ("new" pictures marked as "old")
Psychomotor vigilance task lapse rate | 1-24 hours
  The absolute number of trials in a 5-min test period on which the participant fails to responds with 500ms is calculated as the lapse rate.

SECONDARY OUTCOMES:
fMRI measured neural reactivity (blood oxygen-level dependent signal) | 12-24 hours
  Following sleep or sleep deprivation, regions of interest include amygdala reactivity and connectivity between the amygdala and the ventromedial prefrontal cortex (vmPFC) in response to negative and neutral stimuli.
Heart Rate Reactivity (Beats per minute) | 12-24 hours
  The change in heart rate beats per minute in response to negative and neutral stimuli after sleep or sleep deprivation.
Skin Conductance Reactivity (micro Siemens) | 12-24 hours
  The change in electrodermal activity in response to negative and neutral stimuli after sleep or sleep deprivation.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Cunningham, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Tony Cunningham, Boston, Massachusetts, United States